CLINICAL TRIAL: NCT00096447
Title: A Phase II Evaluation Of Lapatinib (GW572016) (NCI-Supplied Agent, NSC #727989) In The Treatment Of Persistent Or Recurrent Endometrial Carcinoma
Brief Title: Lapatinib in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02631; GOG-0229D; U10CA027469 (NIH); CDR0000393398 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-11-09; First posted 2004-11-10 (Estimated); Results first posted 2015-09-18 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Recurrent Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine

ARMS (1):
- Treatment (lapatinib ditosylate) (Experimental): Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lapatinib ditosylate

INTERVENTIONS:
Drug: lapatinib ditosylate
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb

SUMMARY:
This phase II trial is studying how well lapatinib works in treating patients with recurrent or persistent endometrial cancer. Lapatinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the 6-month progression-free survival of patients with recurrent or persistent endometrial carcinoma treated with lapatinib.

II. Determine the nature and degree of toxicity of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine the objective response rate in patients treated with this drug. II. Determine the duration of progression-free survival and overall survival in patients treated with this drug.

III. Determine the effects of prognostic factors, such as initial performance status and tumor grade, in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral lapatinib once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 22-82 patients will be accrued for this study within 30-67 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial carcinoma

  * Recurrent or persistent disease
  * Histologic confirmation of the original primary tumor is required
* Refractory to curative therapy or standard treatments
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques, including palpation, plain x-ray, CT scan, or MRI OR ≥ 10 mm by spiral CT scan
  * Must have at least 1 target lesion

    * Tumors within a previously irradiated field are considered non-target lesions

      * Disease in an irradiated field as the only site of measurable disease is considered a target lesion provided there has been clear progression of the lesion since the completion of prior radiotherapy
* Must have received 1 prior chemotherapy regimen for endometrial carcinoma

  * Initial therapy may have included high-dose therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment
  * No more than 1 additional prior cytotoxic regimen for recurrent or persistent disease
* Tumor accessible to guided core needle or fine needle biopsy
* Ineligible for a higher priority GOG protocol (e.g., any active GOG phase III protocol for the same patient population)
* Performance status - GOG 0-2 (for patients who have received 1 prior treatment regimen)
* Performance status - GOG 0-1 (for patients who have received 2 prior treatment regimens)
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Cardiac ejection fraction normal by echocardiogram or MUGA
* No gastrointestinal (GI) tract disease resulting in an inability to take oral medication
* No malabsorption syndrome
* No requirement for IV alimentation
* No uncontrolled inflammatory GI disease (e.g., Crohn's or ulcerative colitis)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No sensory or motor neuropathy > grade 1
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to lapatinib
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* At least 4 weeks since prior immunologic agents for the malignant tumor
* No prior trastuzumab (Herceptin^®) or any target-specific therapy directed to the HER family (e.g., gefitinib, erlotinib, or cetuximab)
* At least 6 weeks since prior nitrosoureas or mitomycin for the malignant tumor and recovered
* No prior non-cytotoxic chemotherapy for recurrent or persistent disease
* At least 1 week since prior hormonal therapy for the malignant tumor
* Concurrent hormone replacement therapy allowed
* Recovered from prior radiotherapy
* Recovered from prior surgery
* No prior surgery affecting absorption
* At least 4 weeks since other prior therapy for the malignant tumor
* No prior lapatinib
* No prior anticancer treatment that would preclude study treatment
* Concurrent oral anticoagulants (e.g., warfarin) allowed provided there is increased monitoring of INR
* No concurrent CYP3A4 inducers or inhibitors
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Leslie, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 11/1/2004 and closed to accrual on 9/26/2005.
Groups:
- GW572016: 1500 mg of GW572016 orally every day (cycle = 28 days) until disease progression or adverse effects prohibit further therapy
Period: Overall Study
Arm/Group | GW572016
Started | 31
Completed | 30 (Eligible and treated patients.)
Not Completed | 1
Not completed — Never treated | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients.
Arm/Group | GW572016
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (11.1)
Age, Customized [Number; unit: participants]
  30-39 years | 2
  40-49 years | 4
  50-59 years | 3
  60-69 years | 13
  70-79 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
International Federation of Gynecology and Obstetrics (FIGO) Stage - Recurrent/Persistent [Number; unit: participants] | 30
Histologic Type [Number; unit: participants]
  Adenocarcinoma, Unspecified | 2
  Clear Cell Carcinoma | 3
  Endometrioid Adenocarcinoma | 16
  Mixed Epithelial Carcinoma | 2
  Serous Adenocarcinoma | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Progression-free Survival > 6 Months
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: For those patients whose disease can be evaluated by physical examination, progression was assessed prior to each 28-day cycle. CT scan or MRI if used to follow lesion for measurable disease every other cycle, for up to 5 years.
Population: Eligible and treated patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | GW572016
Number analyzed (Participants) | 30
percentage of participants | 10 [2.3 to 23.9]

2. Primary Outcome: Frequency and Severity of Adverse Events as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) v 3.0
Description: The frequency and severity of all toxicities are tabulated.
Time Frame: Every cycle during treatment and 30 days after the last cycle of therapy.
Population: Eligible and evaluable patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 0: Number of patients who did not experience the specified AE.
- Grade 1 (CTCAE v 3.0): Number of patients who experienced a grade 1 event using Common Terminology Criteria version 3.0
- Grade 2 (CTCAE v 3.0): Number of patients who experienced a grade 2 event using Common Terminology Criteria version 3.0
- Grade 3 (CTCAE v 3.0): Number of patients who experienced a grade 3 event using Common Terminology Criteria version 3.0
- Grade 4 (CTCAE v 3.0): Number of patients who experienced a grade 4 event using Common Terminology Criteria version 3.0
Arm/Group | Grade 0 | Grade 1 (CTCAE v 3.0) | Grade 2 (CTCAE v 3.0) | Grade 3 (CTCAE v 3.0) | Grade 4 (CTCAE v 3.0)
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 30
Participants
  Leukopenia | 29 | 1 | 0 | 0 | 0
  Thrombocytopenia | 28 | 2 | 0 | 0 | 0
  Anemia | 11 | 8 | 10 | 0 | 1
  Cardiovascular | 28 | 1 | 0 | 1 | 0
  Constitutional | 13 | 10 | 7 | 0 | 0
  Dermatologic | 22 | 6 | 1 | 1 | 0
  Gastrointestinal | 5 | 12 | 7 | 6 | 0
  Genitourinary/renal | 29 | 0 | 0 | 1 | 0
  Hemorrhage | 29 | 0 | 0 | 1 | 0
  Lymphatics | 29 | 0 | 1 | 0 | 0
  Musculoskeletal | 27 | 2 | 1 | 0 | 0
  Metabolic | 20 | 5 | 2 | 2 | 1
  Neuropathy | 29 | 1 | 0 | 0 | 0
  Other hematologic | 27 | 3 | 0 | 0 | 0
  Ocular | 26 | 4 | 0 | 0 | 0
  Pain | 25 | 4 | 1 | 0 | 0
  Pulmonary | 27 | 1 | 1 | 1 | 0

3. Secondary Outcome: Percentage of Patients With Tumor Response
Description: Complete and Partial Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.0. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: For those patients whose disease can be evaluated by physical examination, response was assessed prior to each 28-day cycle. CT scan or MRI if used to follow lesion for measurable disease every other cycle, for up to 5 years.
Population: Eligible and treated patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | GW572016
Number analyzed (Participants) | 30
percentage of participants | 3.3 [0.2 to 14.9]

4. Secondary Outcome: Duration of Progression-free Survival
Description: as for outcome 1
Time Frame: Every other cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually for the next 5 years.
Population: Eligible and evaluable patients
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | GW572016
Number analyzed (Participants) | 30
months | 1.82 [1.41 to 3.48]

5. Secondary Outcome: Overall Survival
Description: The observed length of life from entry into the study to death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years.
Population: Eligible and treated patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GW572016
Number analyzed (Participants) | 30
Months | 7.33 [3.94 to 15.77]

6. Secondary Outcome: Prognostic Factors (Performance Status)
Description: Performance status 0 = Fully active, able to carry on all pre-disease performance without restriction.
  Performance status 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature, e.g., light housework, office work.
Time Frame: Baseline
Population: Eligible and evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | GW572016
Number analyzed (Participants) | 30
Participants
  Performance status 0 | 19
  Performance status 1 | 11

7. Secondary Outcome: Prognostic Factor (Histologic Grade)
Description: G1 - Highly differentiated adenomatous carcinoma. G2 - Differentiated adenomatous carcinoma with partly solid areas. G3 - Predominantly solid or entirely undifferentiated carcinoma. Not graded - tumor grade not reported.
Time Frame: Baseline
Population: Eligible and evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | GW572016
Number analyzed (Participants) | 30
Participants
  Grade 1 | 3
  Grade 2 | 6
  Grade 3 | 14
  Not graded | 7

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Also reported are all Serious Adverse Events (SAEs) for up to 5 years after stopping study treatment
Arm/Group | GW572016
Serious Adverse Events (participants affected / at risk) | 10/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GW572016 (N=30)
Hemoglobin (Blood and lymphatic system disorders) | 2
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1
Fistula, Gi - Rectum (Gastrointestinal disorders) | 1
Obstruction, Gi - Jejunum (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 1
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1
Fistula, Gu - Vagina (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GW572016 (N=30)
Rhinitis (Immune system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 2
Leukocytes (Blood and lymphatic system disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 21
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 1
S/N Arrhythmia: Atrial Tachycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 2
Valvular Heart Disease (Cardiac disorders) | 1
Left Venticular Diastolic Dysfunction (Cardiac disorders) | 1
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 2
Hypotension (Cardiac disorders) | 2
Inr (Vascular disorders) | 1
Ptt (Vascular disorders) | 1
Sweating (General disorders) | 3
Weight Gain (General disorders) | 1
Fever (General disorders) | 2
Weight Loss (General disorders) | 3
Rigors/Chills (General disorders) | 1
Fatigue (General disorders) | 20
Insomnia (General disorders) | 6
Nail Changes (Skin and subcutaneous tissue disorders) | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 8
Flushing (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Endocrine disorders) | 2
Diabetes (Endocrine disorders) | 1
Flatulence (Gastrointestinal disorders) | 2
Heartburn (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 1
Distention (Gastrointestinal disorders) | 1
Taste Alteration (Gastrointestinal disorders) | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 1
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 8
Anorexia (Gastrointestinal disorders) | 15
Dehydration (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 15
Diarrhea (Gastrointestinal disorders) | 18
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 1
Hemorrhage, Gu - Vagina (Vascular disorders) | 3
Hemorrhage, Gi - Upper Gi Nos (Vascular disorders) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 1
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1
Inf Unknown Anc: Blood (Infections and infestations) | 1
Infection - Other (Infections and infestations) | 1
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 1
Inf Unknown Anc: Wound (Infections and infestations) | 1
Inf Unknown Anc: Ungual (Nails) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 3
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 1
Edema: Viscera (Blood and lymphatic system disorders) | 1
Edema: Limb (Blood and lymphatic system disorders) | 1
Ast (Metabolism and nutrition disorders) | 2
Proteinuria (Metabolism and nutrition disorders) | 2
Creatinine (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Alt (Metabolism and nutrition disorders) | 2
Alkaline Phosphatase (Metabolism and nutrition disorders) | 6
Bilirubin (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 3
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 1
Mood Alteration - Depression (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Neuropathy-Sensory (Nervous system disorders) | 2
Neuropathy-Motor (Nervous system disorders) | 1
Glaucoma (Eye disorders) | 1
Dry Eye (Eye disorders) | 1
Blurred Vision (Eye disorders) | 3
Pain: Pelvis (General disorders) | 1
Pain: Vagina (General disorders) | 1
Pain: Chest /Thorax Nos (General disorders) | 1
Pain: Chest Wall (General disorders) | 1
Pain: Head/Headache (General disorders) | 2
Pain: Extremity-Limb (General disorders) | 4
Pain: Back (General disorders) | 3
Pain: Joint (General disorders) | 5
Pain: Stomach (General disorders) | 1
Pain: Oral Cavity (General disorders) | 1
Pain: Dental/Teeth/Peridontal (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 5
Pain: Lip (General disorders) | 2
Pain: Middle Ear (General disorders) | 1
Pain: Tumor (General disorders) | 3
Pain: Muscle (General disorders) | 2
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Urinary Retention (Renal and urinary disorders) | 1
Fistula, Gu - Vagina (Renal and urinary disorders) | 1
Fistula, Gu - Genital Tract-Female (Renal and urinary disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 2
Vaginal Discharge (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
The clinical trial was a two-stage design, accruing approximately 25 patients in each stage. Results from a planned interim futility analysis resulted in the early closure of the study. This study stopped early for lack of treatment efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less